CLINICAL TRIAL: NCT06764472
Title: Retrospective Evaluation of a Cohort of Patients Diagnosed With Pre- and Postnatal Urinary Dilatation: Outcome and Long-term Follow-up
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DUCT
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Urinary Tract Dilatation
Keywords: Urinary Tract Dilatation; Children; Ultrasound; Postnatal diagnosis; Prenatal diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective evaluation of a cohort of patients diagnosed with pre- and postnatal urinary dilatation: outcome and long-term follow-up

DETAILED DESCRIPTION:
Urinary tract dilatation is one of the most frequently encountered congenital anomalies in children. Significant improvements in imaging have made it possible to diagnose it earlier, which has led to a major increase in findings during the prenatal period. Before prenatal ultrasound screening became routine, congenital malformations of the kidneys and urinary tract were not diagnosed until they caused symptoms in childhood or occasionally in adult life. Now the vast majority are identified in utero and can be managed prospectively. Antenatal ultrasound diagnosis of urinary tract dilatation is estimated to affect around 1-2% of all pregnancies, and most frequently affects the male sex at a ratio of about 2:12.

The primary goal behind early diagnosis is to be able to monitor the detected abnormalities over time, trying to prevent the onset of possible complications and thus minimize progressive renal damage. However, a disadvantage of this increasing diagnostic accuracy is that it allows the detection of even the smallest of abnormalities, most commonly mild unilateral dilatations of the renal pelvis, which although they have no pathological significance and do not require any kind of intervention, can lead to excessive investigations, unnecessary treatments, and unwarranted anxiety in parents.

The postnatal diagnosis of urinary dilatations not reported on ultrasound scans performed during pregnancy can be traced mainly to three conditions: screening ultrasound scans performed during childhood, kidney and urinary tract monitoring following an intercurrent acute episode such as a urinary tract infection or acute abdominal pain, and follow-up ultrasound scans performed during a hospital stay for another reason.

The presence of urinary tract dilatation can correspond to a spectrum of possible etiologies and underlying nephro-urologic pathologies. In many cases, it is not possible to clarify the underlying etiology of urinary tract dilatation prenatally; rather, it is necessary to wait until the birth and then proceed with in-depth diagnostic investigations based on both first-level imaging methods, such as ultrasonography, and second-level imaging methods, such as micturition cystourethrography (CUM)2 and renal scintigraphy.

Despite the high prevalence, there is still significant variability in the postnatal management of patients diagnosed with urinary dilatation because of the paucity of existing evidence-based correlations between the type of dilatation and the underlying nephro-urologic pathology. This results, in some cases, in the use of unnecessary examinations, which may expose the child to radiation and stress e.g. bladder catheterization for cystography.

The primary aim of this study is to evaluate the diagnostic framing, progression, and different outcomes of patients diagnosed with urinary tract dilatation, considering patients in whom prenatal or postnatal diagnosis was made. The secondary aims are to identify which dilatations are significant, deserving of close follow-up and second-tier examinations (particularly CUM and renal scintigraphy), and to assess the appropriate timing for such examinations, an to assess if the need for postnatal screening is warranted, or whether prenatal screening is sufficient, comparing risk and benefit factors.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients referred to one of the participating centers between January 1 2000 and August 31 2021 for either a prenatal or a postnatal diagnosis of urinary tract dilatation;
* Urinary tract dilatation documented on at least one postnatal ultrasound, with related measurements;
* Presence of at least one other ultrasound performed during follow-up in the postnatal period.

Exclusion Criteria:

* Lack of some of the clinical data considered crucial to the study, particularly incomplete ultrasound reports referable to at least two different ultrasounds performed in follow-up;
* Dilatation with a picture of documented renal lithiasis.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 0-16 years who were referred to the departments and/or outpatient clinics of the participating centers for urinary tract dilataions from January 2000 to August 31 2021. The estimated number of patients to enroll is between 1500 and 2000.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Size parameters | at baseline
  dilatations of the renal pelvis, renal calices and ureter
Presence of hyperecogenicity | at baseline
  yes/no
Presence of renal and/or bladder abnormalities | at baseline
  yes/no
Polar diameter of the kidneys | at baseline
  mm

CONTACTS AND LOCATIONS:
Overall Officials: Claudio La Scola, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy